CLINICAL TRIAL: NCT05781776
Title: Comparison of Effects of Otago Exercise Program vs. Gaze Stability Exercise on Balance and Fear of Fall in Older Adults
Brief Title: Otago Exercise Program And Gaze Stability Exercise In Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MSECO4/2019
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Balance
Keywords: Berg balance scale; Fall efficacy scale-International; Rehabilitation; Exercises; Older Adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Two arms pretest-posttest design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago exercise program group (Experimental): Participants performed Otago exercise program and core muscle strengthening exercises for eight weeks (thrice a week).
  Interventions: Other: Otago exercises and core strengthening
- Gaze stability exercises group (Active Comparator): Participants performed Gaze stability exercises and core muscle strengthening exercises for eight weeks (thrice a week).
  Interventions: Other: Gaze stability exercises and core strengthening

INTERVENTIONS:
Other: Otago exercises and core strengthening — Otago exercise program consisted of strengthening and balance exercises. The strengthening exercises focus on major lower limb muscles. Progression of exercises was done by increasing the duration and then intensity.
  Balance exercises involved knee bends, backward walking, walking, and turning around, sideways walking, tandem stance (heel to toe), tandem walk (heal to toe walk), one leg stand, heel walking, toe walk, heel to toe walking backward, sit to stand and stair walking. Balance exercises progressed with varying levels of support depending on their balance and confidence. The individuals repeated each exercise 10 times.
  Arms: Otago exercise program group
Other: Gaze stability exercises and core strengthening — The exercise protocol in Gaze Stability exercises included adaptation exercises and substitution exercises. In adaptation exercises, individuals performed rapid, active head rotations while watched a visual target with the target remaining stationary. Substitution exercises, individual performed eye-head movements between targets with the goal of seeing clearly during the task. That target moved in the opposite direction of head movement.
  Adaptation exercises included: Horizontal and vertical (stationary target) viewing exercises done with a near target, sitting. Horizontal and vertical (stationary target) viewing exercises done with near and far targets (6-10 feet), sitting. Horizontal and vertical (stationary target) viewing exercises were done with near and far targets, standing.
  Arms: Gaze stability exercises group

SUMMARY:
Fall occurrences and the associated risk of injury are debilitating and major health concerns in the older population. Several interventions have been investigated and implemented to address the needs of balance impairments and to reduce the increased risk of falls. This study aimed to compare the effectiveness of the Otago exercise program (OEP) and gaze stability exercises (GSE) on balance and the risk of falls in older adults residing at an old age home facility. 30 elderly participants were equally and randomly divided into two groups: Group OEP received the OEP and group GSE received GSE for eight weeks (thrice a week). In addition, both groups also performed core muscle-strengthening exercises. The Berg balance scale (BBS) and the Fall efficacy scale-International (FES-I) were the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Participants were independent in ambulation
* They were performing activities of daily living independently
* They had impaired balance having Berg Balance Scale (BBS) score between 35-45
* They had dynamic Gait Index score between 11-19
* They had mini-mental status exam scores > 22

Exclusion Criteria:

* severe vision or hearing impairment,
* neurological disorders including epilepsy, Alzheimer's disease, vertigo, Parkinson's disease, etc.,
* muscular disorders which limit functional activity (Osteoarthritis, Rheumatoid arthritis, etc.),
* taking medications that affect balance,
* severe cardiovascular conditions,
* recent Lower limb injury or Surgery,
* obesity

Ages: 65 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | 8 weeks.
  This tool encompasses both static and dynamic balance components across 14 different activities (5 static and 9 dynamic) performed by the patient graded on varying difficulty levels for different balance conditions (sitting balance, standing up, turning around, walking on an even surface, walking on steps, and while changing body position). The BBS utilizes an ordinal grading on a 5-point scale (0-4) to rate the 14 task items, producing a global score of 56 with the lower score assigned to poor performance (score-0) and a greater score representing the better outcomes (score-4).
Fall efficacy Scale- International (FES-I) | 8 weeks.
  The FES-I form consists of 16 items related to various functional activities. The participant is asked to rate the level of each activity on a 4-point Likert scale. A higher score implies a greater fear of falls and lower score imply better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th., Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kp N, D A, Nawed A, Nuhmani S, Khan M, Alghadir AH. Comparison of effects of Otago exercise program vs gaze stability exercise on balance and fear of fall in older adults: A randomized trial. Medicine (Baltimore). 2024 Jun 7;103(23):e38345. doi: 10.1097/MD.0000000000038345. PMID 38847714